CLINICAL TRIAL: NCT06571955
Title: Anterior Cruciate Ligament (ACL) Reconstruction with a New Generation of LARS Artificial Ligament
Brief Title: ACL Reconstruction with a New Generation of LARS Artificial Ligament
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MOVMEDIX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD/PT.03
Record Dates: First submitted 2024-07-15; First posted 2024-08-26 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: ACL Injury
Keywords: ACL; Artificial ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LARS grafted (Experimental): Patients implanted with grafted ligament (new generation)
  Interventions: Device: Implantation of LARS artificial grafted ligament to treat ACL injury
- Control (Active Comparator): Patients implanted with non-grafted ligament (current generation)
  Interventions: Device: Implantation of LARS artificial non-grafted ligament to treat ACL injury

INTERVENTIONS:
Device: Implantation of LARS artificial grafted ligament to treat ACL injury — Implantation procedure will be realized by a well-trained orthopaedic surgeon and will consist of ACL repair using LARS artificial grafted ligament.
  Arms: LARS grafted
Device: Implantation of LARS artificial non-grafted ligament to treat ACL injury — Implantation procedure will be realized by a well-trained orthopaedic surgeon and will consist of ACL repair using LARS artificial non-grafted ligaments.
  Arms: Control

SUMMARY:
This clinical investigation is intended to demonstrate the safety of the new generation of LARS ligaments and compare this new generation (grafted ligament) of artificial ligament to the LARS current artificial ligament (non-grafted ligament) which is CE marked since 1997, in case of ACL injury. The new generation of LARS artificial ligament is expected to improve physiological response by enhancing fibroblast proliferation, fibroblast organization and collagen type I & III secretion. This physiological response leads to a better osseo-integration of the ligaments. Therefore, the study is expected to demonstrate the investigational device safety and biomechanical improvements.

DETAILED DESCRIPTION:
Forty subjects over 40 years old with acute ACL injury will be included. A follow-up program is planned over 1 year per subject (days 7, 15, 30, 60, 90, 180, 365) based on physical therapy, biological analysis and biomechanical measurements.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the grafted ligament
* Subject provides written informed consent approved by the Ethics Committee prior to any clinical investigation related procedure
* Subject must agree to undergo all clinical investigation plan - required clinical follow-up visits
* Subject must agree not to participate in any other clinical investigation for a period of 1 year following the procedure
* Male and female subjects over 40 years old
* MRI positive for full acute ACL injury
* Arthrometric evaluation (KT1000) with a side-to-side difference greater than 3 mm
* Symptomatic subjects with no previous knee injury
* Subjects without concomitant pathologies (fracture, infections, immunodepression, HIV, HCV) that could influence the outcome of the study or prevent the subject from following the post-operative follow-up program as per protocol
* I and II degree chondral lesions

Exclusion Criteria:

* Subjects under 40 years old
* III and IV degree chondral lesions
* Associated ligament injuries
* Meniscus suture (e.g. hndle bucket meniscal tears) that compromise the rehabilitation program
* History for sepsis
* Subjects with concomitant pathologies (fracture, infections, immunodepression, HIV, HCV,) that could influence the outcome of the study or prevent the subject from following the post-operative follow-up program as per protocol
* Previous knee injuries
* Septic arthritis
* Infected tissues
* Pregnancy
* Overweighed, obese subject (>100kg)
* History of metabolic bone disease
* Inflammatory joint disease
* Known neoplastic disease
* Medical treatment (e.g steroid)
* HIV positive subject
* Hepatitis positive subject
* Allergy to Titanium, PET, Ugurol, Gentamicin, Polystyrene Sulfonate, other medication

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Device Effect (SADE) | 6 months
  Primary outcome will evaluate the safety of the grafted ligament by reporting the number of SADE(s) in the Experimental Arm.

SECONDARY OUTCOMES:
Assessment of patients' opinion about their knee and associated problems | 12 months
  Patient will answer the questionnaire KOOS (Knee Injury and Osteoarthritis Outcome Score) pre-surgery, 90, 180 and 365 days post-surgery.
  This is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems both on short-term and long-term. The KOOS questionnaire includes five dimensions that are relevant to patients: pain, symptoms, daily activities, sports and recreation, and quality of life. Each of these dimensions is scored separately, using a Likert scale with five possible answers ranging from 0 (no problems) to 4 (extreme problems). The scores for each dimension are calculated by summing the answers to the relevant questions. The resulting scores are then transformed to a scale from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problems. Answers to the questionnaire pre-surgery will be compared to the answers collected at 90, 180 and 365 days post-surgery.
Assessment of patients' pain intensity | 12 months
  The Visual Analogue Scale (VAS) will be used to measure the intensity or frequency of various symptoms, most commonly pain. Patients will be asked to mark a point on the line that represents their perception of their current state pre-surgery, 90, 180 and 365 days post-surgery. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Scores obtained pre-surgery will be compared to the scores obtained at 90, 180 and 365 days post-surgery.
Assessment of overall knee function | 12 months
  The IKDC Subjective Knee Evaluation Form is used to evaluate the knee. The questionnaire looks at 3 categories: symptoms, sports activity and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. The sports activity subscale focuses on functions such as; going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks patients 1 simple question - how is their knee at present versus how was their knee prior to injury.
  Scores are obtained by summing the individual items and then transforming the crude total to a scaled number that ranges from 0 to 100. Higher scores indicate higher levels of function and lower levels of symptoms. Patients will complete the IKDC form pre-surgery, 90, 180 and 365 days post-surgery. Scores obtained pre-surgery will be compared to the scores obtained at 90, 180 and 365 days post-surgery.
Assessment of posterior-anterior knee laxity | 12 months
  Posterior-anterior knee laxity is measured using a KT-1000 arthrometer. The subject lies in a supine position with the knee flexed about 20°, a support is placed below the knee proximal to the popliteal space. The subject is told to relax in this position. The arthrometer is then placed above the tibia and attached firmly by two bands. After adjusting the zero, the tibia is pulled anteriorly using the handle on the arthrometer. An audible indication will be noticed at 15, 20 and 30 pounds (approx. 6, 9 and 13kg) of force. Moreover, a manual maximum measure is performed pulling the tibia with a hand on the back of the shank, until the foot is raised. Displacement is measured in millimeters and compared with the healthy leg measurements. The difference between the legs should be 1mm - 15mm.
  Knee laxity will be measured pre-surgery, 45, 90, 180 and 365 days post-surgery. Values at pre-surgery will be compared to the ones from post-surgery mesurements.
Assessment of knee flexors-extensors strength | 12 months
  Knee flexors-extensors strength assessment will be measured using an Isokinetic machine and superficial EMG evaluation. The subject performs an isokinetic concentric evaluation with a fixed velocity of 90°/s with a range of motion of 0-90° of knee flexion. After warming-up, subject is asked to sit on the resting chair of the dynamometer, the subject is then secured with body straps. The starting position is 90° flexion for the knee and 90° for the hip joint. The subject is instructed to extend the knee till 0° flexion and then to flex the knee back at 90° with maximum exertion. The test is performed firstly on the healthy side and then on the injured side. Peak forces are compared between the legs.
  Knee flexors-extensors strength will be measured pre-surgery, 90, 180 and 365 days post-surgery. Values at pre-surgery will be compared to the ones from post-surgery mesurements.
Assessment of stabilometry | 12 months
  The subject is asked to stay still on a force platform for 10 seconds, firstly standing only on one leg with the arms folded across the chest. The test is then repeated on the other leg. The motion/change of the centre of pressure is used to quantify ellipse area to measure stability. Usually, ellipse area results for stabilometry test show differences between the healthy and the injured leg.
  Stabilometry will be measured in both legs pre-surgery, 45, 90, 180 and 365 days post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guliano Cerulli, MD, Principal Investigator — Instituto di Ricerca Traslazionale Per l'Apparato Locomotore Nicola Cerulli (I.R.T.A.L)
Locations (1):
- Instituto di Ricerca Traslazionale Per l'Apparato Locomotore Nicola Cerulli (I.R.T.A.L), Perugia, Italy

IPD SHARING:
Plan to Share IPD: No